CLINICAL TRIAL: NCT04602650
Title: Microbial Determinants of Dementia Risk in Type 2 Diabetics of Mexican Descent
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0201
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal bacterial DNA specimens will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 Diabetic: Type 2 diabetic individuals of Mexican descent.
- Non-diabetic Controls: Non-diabetic individuals of Mexican descent.

SUMMARY:
Type 2 diabetes (T2D) predisposes individuals to neurodegeneration and dementia, including Alzheimer's Disease (AD); yet the link between metabolic and neurodegenerative disorders remains unknown. Here, the investigators will study a well-defined human population with increased prevalence and early onset of both T2D and AD, individuals of Mexican descent living in South Texas. The study will begin to explore the possibility that disruption of the structure of the bacterial community residing in the gut in type 2 diabetic individuals of Mexican descent living in South Texas is directly related to the increased prevalence of early onset AD in this population. In this study, the investigators will perform gene sequencing on DNA isolated from fecal samples to identify and compare the populations of bacteria living in individuals with T2D versus non-diabetic controls. The investigators will analyze the findings to determine if the community structure of the gut microbiome of individuals of Mexican descent with T2D is significantly altered compared to that of non-diabetics within the same population. The investigators' findings could lead to the identification of early indicators of dementia onset as well as novel therapies for treating metabolic and neurodegenerative diseases.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) as a common antecedent of pathological neurodegeneration and dementia, including Alzheimer's Disease (AD); yet the mechanistic link between metabolic and neurodegenerative disorders remains unresolved. Here, the investigators will study a well-defined human population with increased prevalence and early onset of both T2D and AD, individuals of Mexican descent living in South Texas. The study will lay critical groundwork toward addressing the investigators' overarching hypothesis that dysbiosis of the gut microbiome in type 2 diabetic individuals of Mexican descent living in South Texas is causally related to the increased prevalence of comorbid, early onset AD in this population. In this study, the investigators will perform state-of-the-art metagenomic 16S ribosomal RNA (rNRA) gene sequencing and bioinformatic analysis on fecal samples collected from type 2 diabetic and non-diabetic control individuals of Mexican descent to test the working hypothesis that the community structure of the gut microbiome of individuals of Mexican descent with T2D is significantly altered compared to that of nondiabetics within the same population. To the investigators' knowledge, this multidisciplinary pilot study will be the first to investigate the gut microbial community structure of type 2 diabetic versus that of nondiabetic individuals of Mexican descent. Furthermore, it has the potential to provide mechanistic insight into how T2D predisposes individuals to the neuropathology and cognitive impairment characteristic of AD and to identify a novel class of interventions that target the host gut microbiome for the prevention of early onset AD in a predisposed population, as well as the population at large.

Human subjects will be recruited through the University of Texas Medical Branch at Galveston (UTMB) Endocrinology and pre-screened to confirm that the potential participants meet established inclusion and exclusion criteria as either T2D or nondiabetic controls, as defined in the UTMB human subjects protocol associated with this project. Pre-screened participants that meet the defined criteria will be invited to attend an appointment with a study coordinator held at the UTMB Clinical Research Center. Consented and enrolled study participants will be asked to complete medical history, dietary preference, and gastrointestinal function questionnaires and instructed as to how to use the provided OMNIgene-GUT RNA (OMR)-200 fecal sample collection kit (DNA GenoTek). Participants will submit the collected fecal sample via shipment of a pre-paid and labeled shipping envelope. Samples will be deidentified and stored at -80oC in the Buffington Lab prior to shipment to the Baylor College of Medicine Center for Metagenomic and Microbiome Research (CMMR) for metagenomic 16S rRNA gene sequencing. Briefly, bacterial genomic DNA will be extracted using the MagAttract PowerSoil Kit (Qiagen) and the 16S ribosomal DNA (rDNA) V4 region will be amplified by polymerase chain reaction (PCR) and sequenced on the MiSeq platform (Illumina). 16S rRNA gene read pairs will be demultiplexed based on unique molecular barcodes added to primers used for amplification and reads will be merged using USEARCH. 16S rRNA gene sequences will be clustered into Operational Taxonomic Units (OTUs) using the UPARSE algorithm and mapped to an optimized version of the SILVA database to determine taxonomies. The investigators will then use a custom script developed by the CMMR to construct a rarefied OTU table for downstream analyses of alpha-diversity, beta-diversity, and phylogenetic trends to identify any changes in community structure between type 2 diabetic and non-diabetic individuals of Mexican descent enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

Type 2 Diabetic Inclusion Criteria

1. Male or female with a diagnosis of type 2 diabetes.
2. Ages 50 to 70 years.
3. Mexican descent living in Texas.
4. Participant is willing and able to give informed consent for participation in the study.

Non-Diabetic Control Inclusion Criteria

1. Male or female without history of type 2 diabetes.
2. Ages 50 to 70 years.
3. Mexican descent living in Texas.
4. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

Type 2 Diabetic Exclusion Criteria

1. Hypertension that is not controlled by greater than 2 medications.
2. Chronic kidney disease, CKD greater than 3.
3. History of coronary bypass or stint placement.
4. Current pregnancy.
5. Subjects with a history of inflammatory bowel disease, Celiac disease or active diverticular disease.
6. Other medical condition or medication administration deemed exclusionary by the study investigators.

Non-Diabetic Control Exclusion Criteria

1. Hypertension that is not controlled by greater than 2 medications.
2. Chronic kidney disease, CKD greater than 3.
3. History of coronary bypass or stint placement.
4. Current pregnancy.
5. Subjects with a history of inflammatory bowel disease, Celiac disease or active diverticular disease.
6. Other medical condition or medication administration deemed exclusionary by the study investigators.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will study subjects of Mexican descent living in Texas (aged 50-70 years) with a history of type 2 diabetes (T2D) (n=50, anticipated) and non-diabetic controls (aged 50 - 70 years) (n=50, anticipated).
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Fecal Microbial Gene Sequencing | Baseline
  Metagenomic 16S ribosomal RNA (rRNA) gene sequencing will be performed on subject samples to determine the presence and measure the relative abundance of operational taxonomic units representative of bacterial genera, species, and strains present in the fecal sample.

SECONDARY OUTCOMES:
Gastrointestinal health as measured by gastrointestinal symptom rating scale | Baseline
  The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort). The sum of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 15 (best outcome) to 105 (worst outcome). GSRS will be measured at baseline.
Food Preference Questionnaire | Baseline
  The Food Preference Questionnaire (FPQ) is a specific 3-item questionnaire. Subjects are asked to first indicate whether they identify as vegan, vegetarian, pescetarian, or none of the above. They are then asked whether they have any food allergies to eleven common food allergies and have the option to specify a food allergy not listed under "Other." Finally, the subject is asked to indicate preference (ranging from "dislike a lot" to "like a lot") for 59 specific food items in a table. FPQ will be acquired at baseline.
  [Modified from "Food Preference Questionnaire for Adolescents and Adults," University College London, Institute of Epidemiology and Health Care, Research Department of Behavioural Science and Health.]
Neurological History Questionnaire | Baseline
  The Neurological History Questionnaire (NHQ) is a specific 2-item questionnaire. First, subjects are asked to indicate whether they have ever been diagnosed one of ten common neurological disorders. In the second question, subjects are asked to indicate whether they have experienced either of the following neurological events: (1) ischemic stroke or (2) mild traumatic brain injury.

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Buffington, PhD, Principal Investigator — University of Texas Medical Branch Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Matz LM, Shah NS, Porterfield L, Stuyck OM, Jochum MD, Kayed R, Taglialatela G, Urban RJ, Buffington SA. Gut pathobiont enrichment observed in a population predisposed to dementia, type 2 diabetics of Mexican descent living in South Texas. Front Microbiomes. 2024;3:10.3389/frmbi.2024.1456642. doi: 10.3389/frmbi.2024.1456642. Epub 2024 Dec 3. PMID 40969174